CLINICAL TRIAL: NCT03960021
Title: Immune Mechanisms After Radiofrequency Ablation of Pulmonary Metastases From Colorectal Cancer Origin- ARFIM Study
Brief Title: Immune Mechanisms After Radiofrequency Ablation of Pulmonary Metastases From Colorectal Cancer Origin
Acronym: ARFIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Bergonié (Other)
Collaborators: Groupement Interrégional de Recherche Clinique et d'Innovation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IB 2018-03; 2018-A01996-49 (Other: ID-RCB ANSM)
Record Dates: First submitted 2019-04-02; First posted 2019-05-22 (Actual); Results first posted 2025-10-24 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-09

CONDITIONS: Immune Evasion, Tumor; Neoplastic Cells, Circulating; Circulating Tumor Cell; Pulmonary Metastasis; Colo-rectal Cancer
Keywords: Colo-rectal cancer; Lung metastasis; Radiofrequency ablation; Tumor infiltrating lymphocytes; Circulating tumor cells; Circulating DNA
MeSH Terms: conditions — Neoplasms; Neoplastic Cells, Circulating; Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): Each patient is treated with 2 RFA interventions.
  Interventions: Radiation: RFA interventions

INTERVENTIONS:
Radiation: RFA interventions — Each patient is treated with 2 RFA interventions. Abiopsy of one metastasis is done at each RF session. Histological samples are sent to the Bio-pathology department of Institut Bergonié for tumor infiltrating lymphocytes counting. Primary outcome results from this counting (stromal TILs ≥ 20% is considered as a significant level, a comparative measurement before and after RF will be performed). In parallel blood samples are performed before and after RFA to analyze the kinetics of peripheral blood T lymphocytes subsets, tumoral circulating cells and tumoral DNA.

SUMMARY:
Local percutaneous thermal ablation is frequently proposed in the management of metastatic diseases. Radiofrequency ablation (RFA) has demonstrated good results when the metastatic disease is limited and slowly evolving. The destruction of solid metastasis by RF leads to inflammatory and immunological mechanisms that remain poorly understood. These pathological events may influence the overall and anti-tumor host immune responses. The purpose of the study is to identify and quantify some immune mechanisms triggered by RFA of pulmonary metastases from colorectal cancer origin.

DETAILED DESCRIPTION:
RFA could provide activatory signals and become a source of tumor antigens for the immune system. Generating a massive and transient release of antigens, RFA could boost lymphocyte proliferation and production of inflammatory cytokines in response to tumor extracts. Herein, the investigator aims to demonstrate that RFA can amplify the specific T cell response in metastatic cancer patients. In order to ensure this, he plans to assess and quantify tumor infiltrating lymphocytes through tumoral biopsies. He also plans to measure the CD4, CD8 and NK lymphocytes release, the circulating DNA and tumoral cells release, during RFA of lung metastases. On tumoral biopsies, the expression of PDL-1 ligand will also be evaluated and measured. Participants with bilateral metastases or with 5 or more unilateral metastases will be recruited. The two RFA interventions will be carried out within 4-6 weeks of each other. Blood samples and tumoral biopsies will be performed during each intervention. Biopsies will be performed on a metastasis before the thermal ablation. Blood samples will be performed just before RFA, 30 min after RFA and one day after. Analysis, identification and measure of lymphocytes release will be performed with flow cytometry. All analysis and measurements will be performed in the Bio-Pathology department of Institut Bergonié.

ELIGIBILITY:
Inclusion Criteria:

1. Patient older than 18 years-old.
2. OMS performance status ≤ 2.
3. Colorectal cancer histologically established previously.
4. Primary tumor resected.
5. Lung metastasis:

   1. Bilateral metastasis (or unilateral metastases that need to undergo the RF in two separate sessions due to the number of metastases ≥ 5)
   2. Maximal diameter ≤ 4 cm,
   3. non or slowly progressive, with or without chemotherapy,
   4. eligible to RFA.
6. Thorax-abdomen-pelvis CT scan and PET scan:

   1. performed within 8 weeks before inclusion
   2. finding no more than 10 metastatic nodules (liver + lung or lung alone)
7. Maximum of 8 weeks between the last cycle of chemotherapy and the first RFA.
8. Decision of local treatment agreed at the multidisciplinary digestive tumor board.
9. Life expectancy ≥ 3 months.
10. Voluntarily signed and dated written informed consent prior to any study specific procedure.
11. Patients with a French social security in compliance with the Law relating to biomedical research (Article 1121-11 of French Public Health Code).

Exclusion Criteria:

1. Other than lung or liver metastases.
2. Contraindication to general anesthesia.
3. Contraindication to RFA: tumor location (< 1cm from the hilum), lung insufficiency (FEV/sec < 1l),
4. Pregnant or lactating women.
5. Concomitant participation to another interventional research.
6. Patient unable to follow and comply with the study procedures because of any geographical, social or psychological reasons.
7. Patient deprived of liberty or under legal protection measure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2022-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean PALUSSIERE, MD, Principal Investigator — Institut Bergonié
Locations (1):
- Institut Bergonie, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miles J, Soubeyran I, Marliot F, Pangon N, Italiano A, Bellera C, Ward SG, Pages F, Palussiere J, Larijani B. Determination of Interactive States of Immune Checkpoint Regulators in Lung Metastases after Radiofrequency Ablation. Cancers (Basel). 2022 Nov 22;14(23):5738. doi: 10.3390/cancers14235738. PMID 36497220

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single arm
Started | 20
Completed | 17
Not Completed | 3
Not completed — did not undergo the 2 radiofrequency ablations. | 3

BASELINE CHARACTERISTICS:
Arm/Group | Single arm
Number analyzed (Participants) | 17
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 70.8 [68.3 to 76.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 17

OUTCOME MEASURES:

1. Primary Outcome: Immune Response Triggered by RFA: Change From Rate of Tumor Infiltrating T Lymphocytes on Tumoral Stroma Measured Before and After RFA1.
Time Frame: Day 1
Population: Biological analyses could not be performed (technical reasons related to the machine). As such, it was not possible to assess this outcome and report summary statistics as expected.
  No attempt will be made in the future to collect and/or report the data
Arm/Group | Single arm
Number analyzed (Participants) | 0

2. Primary Outcome: Immune Response Triggered by RFA: Change From Rate of Tumor Infiltrating T Lymphocytes on Tumoral Stroma Measured Before and After RFA2.
Time Frame: Week 6
Population: as for outcome 1
Arm/Group | Single arm
Number analyzed (Participants) | 0

3. Primary Outcome: Immune Response Triggered by RFA: Quantification of Interaction of PD-1 and PD-L1 in Lung Metastases Using Immune Förster Resonance Energy Transfer (iFRET).
Time Frame: Day 1
Population: as for outcome 1
Arm/Group | Single arm
Number analyzed (Participants) | 0

4. Primary Outcome: Immune Response Triggered by RFA: Quantification of Interaction of PD-1 and PD-L1 in Lung Metastases Using Immune Förster Resonance Energy Transfer (iFRET).
Time Frame: Week 6
Population: as for outcome 1
Arm/Group | Single arm
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year after radiofrequency ablation
Arm/Group | Single arm
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 19/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single arm (N=20)
Vomiting (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 2 (2)
Pain (General disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 19 (37)
Respiratory; thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Vascular disorders - Other (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-10): https://cdn.clinicaltrials.gov/large-docs/21/NCT03960021/Prot_SAP_000.pdf